CLINICAL TRIAL: NCT03346109
Title: Prospective Randomised Controlled Non-inferior Trial Studying the Feasibility and Potential Quality of Life Benefits of Medial Group Retropharyngeal Node Sparing in Nasopharyngeal Carcinoma
Brief Title: To Study the Feasibility and Quality of Life of Medial Group Retropharyngeal Node Sparing in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-FXY-114
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; medial group retropharyngeal node
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRLN sparing group (Experimental): Patients in medial group retropharyngeal node（MRLN） sparing group will not routinely receive MRLN irradiation to 56Gy/33Fr
  Interventions: Radiation: medial group retropharyngeal node（MRLN） sparing
- MRLN prophylactic irradiation group (No Intervention): Patients in MRLN prophylactic irradiation group will always receive MRLN irradiation to 56Gy/33Fr

INTERVENTIONS:
Radiation: medial group retropharyngeal node（MRLN） sparing — Patients in MRLN sparing group will not routinely receive MRLN irradiation; while patients in MRLN prophylactic irradiation group will always receive MRLN irradiation to 56Gy/33Fr.
  Arms: MRLN sparing group

SUMMARY:
This is an randomized, controlled, phase 3 clinical trial. The purpose of this study is to evaluate whether medial group retropharyngeal node （MRLN） sparing could reduce the incidence of radiation-caused dysphagia and improve patients' quality of life without compromising survival rate.

DETAILED DESCRIPTION:
In this study, patients with non-keratinizing stage T1-4 N0-3 M0 NPC(UICC/AJCC 8th edition), except for patients with MRLN metastasis, are randomly assigned to receive MRLN sparing or prophylactic irradiation . Patients in MRLN sparing group will not routinely receive MRLN irradiation to 56Gy/33Fr; while patients in MRLN prophylactic irradiation group will always receive MRLN irradiation to 56Gy/33Fr. Our primary endpoint is local relapse-free survival (LRFS). Secondary end points include overall survival (OS), incidence of out-field recurrence rate, toxic effects, and quality of life (QOL).All efficacy analyses are conducted in the intention-to treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients without medial group retropharyngeal node metastasis;
2. Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type);
3. Tumor staged as T1-4N0-3(according to the 8th AJCC edition);
4. No evidence of distant metastasis (M0);
5. Satisfactory performance status: Karnofsky scale (KPS) ≥ 70;
6. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Patients with medial group retropharyngeal node metastasis;
2. Aged > 65 or < 18;
3. Treatment with palliative intent;
4. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer;
5. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period);
6. With history of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume);
7. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes;
8. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Local replase-free survival rate | 3 Year
  Local failure-free survival is calculated from randomization to the first local failure

SECONDARY OUTCOMES:
Incidence of acute and late toxicity | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Incidence of out-field recurrence rate | 3 Year
  Number of participants with out-field recurrence
Dysphagia related quality of life | 1 year
  Quality of life (QOL) as assessed by EORTC quality of life questionnaire(QLQ)-HN35
Overall survival | 3 Year
  Overall survival is calculated from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mao YP, Wang SX, Gao TS, Zhang N, Liang XY, Xie FY, Zhang Y, Zhou GQ, Guo R, Luo WJ, Li YJ, Liang SQ, Lin L, Li WF, Liu X, Xu C, Chen YP, Lv JW, Huang SH, Liu LZ, Li JB, Tang LL, Chen L, Sun Y, Ma J. Medial retropharyngeal nodal region sparing radiotherapy versus standard radiotherapy in patients with nasopharyngeal carcinoma: open label, non-inferiority, multicentre, randomised, phase 3 trial. BMJ. 2023 Feb 6;380:e072133. doi: 10.1136/bmj-2022-072133. PMID 36746459